CLINICAL TRIAL: NCT03369808
Title: Immunogenicity And Safety Of An Alum-Adjuvanted Inactivated H7N9 Influenza Vaccine
Brief Title: A Clinical Trail Of An Adjuvanted Inactivated H7N9 Influenza Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016L09902
Record Dates: First submitted 2017-11-22; First posted 2017-12-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: H7N9 Influenza
Keywords: H7N9

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 7.5μg H7N9 Vaccine (Experimental): Participants will receive 2 doses of 7.5μg hemagglutinin antigen of H7N9 vaccine at 21-day intervals.
  Interventions: Biological: 7.5μg H7N9 Vaccine
- 15μg H7N9 Vaccine (Experimental): Participants will receive 2 doses of 15μg hemagglutinin antigen of H7N9 vaccine at 21-day intervals.
  Interventions: Biological: 15μg H7N9 Vaccine
- 30μg H7N9 vaccine (Experimental): Participants will receive 2 doses of 30μg hemagglutinin antigen of H7N9 vaccine at 21-day intervals.
  Interventions: Biological: 30μg H7N9 Vaccine
- Aluminum hydroxide adjuvant (Placebo Comparator): Participants will receive 2 doses of aluminum hydroxide adjuvant at 21-day intervals.
  Interventions: Biological: Aluminum Hydroxide Adjuvant
- Phosphate buffer solution (Placebo Comparator): Participants will receive 2 doses of phosphate buffer solution at 21-day intervals.
  Interventions: Biological: Phosphate Buffer Solution

INTERVENTIONS:
Biological: 7.5μg H7N9 Vaccine — The vaccine was a inactivated, whole virion preparation of the influenza A/Shanghai/2/2013(H7N9) virus, propagated in embryonated chicken eggs，mixed with aluminum hydroxide adjuvant.
  Arms: 7.5μg H7N9 Vaccine
Biological: Phosphate Buffer Solution — 0.5ml phosphate buffer solution
  Arms: Phosphate buffer solution
Biological: Aluminum Hydroxide Adjuvant — 0.5ml aluminum hydroxide adjuvant
  Arms: Aluminum hydroxide adjuvant
Biological: 15μg H7N9 Vaccine — The vaccine was a inactivated, whole virion preparation of the influenza A/Shanghai/2/2013(H7N9) virus, propagated in embryonated chicken eggs，mixed with aluminum hydroxide adjuvant.
  Arms: 15μg H7N9 Vaccine
Biological: 30μg H7N9 Vaccine — The vaccine was a inactivated, whole virion preparation of the influenza A/Shanghai/2/2013(H7N9) virus, propagated in embryonated chicken eggs，mixed with aluminum hydroxide adjuvant.
  Arms: 30μg H7N9 vaccine

SUMMARY:
The aim of this study is to investigate the immunogenicity and safety of the inactivated whole-virion vaccine for teenagers and adults.

The investigators will test the vaccine in participants aged 12-60 years, for a randomized, blind, placebo-controlled, age-stratified clinical study. The investigators designed three dosage groups: 7.5 μg,15 μg and 30 μg of hemagglutinin antigen. According to the age of the subjects, Each group was divided into different age subgroups. Phosphate buffer solution and Aluminum hydroxide adjuvant as placebo controls were both set up in the subgroups.Participants will receive 2 doses of vaccine at 21-day intervals.Safety up to 6 months and changes in hemagglutinin inhibition (HI) titers at 21 days after each vaccination were determined.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 12 years,healthy population
* Subjects/ (and the guardian) informed consent, voluntarily participated and signed the informed consent form, with the ability to use thermometers, scales and to fill in diary cards as required
* To comply with the requirements of clinical trial program, receive blood test before and after immunization and cooperate with follow-up

Exclusion Criteria:

* A history of influenza A (H7N9) virus infection or suspected infection Abnormal blood routine, blood biochemistry and urine routine examination indexes
* Allergy to any component in the vaccine (allergy history of any previous vaccination), especially for egg allergy
* History of asthma, history of thyroid resection, vascular nerve edema, diabetes mellitus, hypertension can not be controlled by medicine, liver and kidney diseases or malignant tumor history
* Suffered from any serious illness, such as cancer, autoimmune disease, progressive atherosclerotic disease or complications of diabetes, chronic obstructive pulmonary disease, need oxygen therapy for acute or progressive liver or kidney disease, congestive heart-failure etc.
* History of signs disease or symptoms of neurological symptoms
* Suffering from severe chronic diseases (such as Down's syndrome, diabetes, sicklemia or neurological disorders, Green's Barre syndrome)
* Acute attacks of various acute or chronic diseases in the past 7 days
* Known or suspected of respiratory disease, acute infection or chronic disease active period, HIV infection, cardiovascular disease, severe hypertension, malignant tumor during treatment, skin diseases
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition etc
* No spleen, functional absence of spleen, and splenectomy or splenectomy without any condition
* Autoimmune diseases or immunodeficiency have been treated with immunosuppressive agents in the past 6 months
* History of epilepsy, convulsions, or a family history of psychosis
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities), or obvious bruising or coagulopathy
* The blood products were received within 3 months prior to the acceptance of the vaccine
* Received a live vaccine within 14 days prior to receiving the vaccine, or received a subunit or inactivated vaccine within 7 days
* Fever within 3 days prior to vaccination, axillary temperature ≥38 ℃
* Being febrile When inoculating vaccine, axillary temperature >37.0 ℃
* Women are pregnant or in the near future planned pregnancy or pregnancy test positive
* Participants in another clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Reactogenicity Events | Continuous observation for 30 days after two inoculations
  * For each group the incidence rate of subjects with solicited AE(s) with 95% confidence interval
  * For each group the incidence rate of subjects with solicited SAE(s) with 95% confidence interval

SECONDARY OUTCOMES:
Number of participants that presented seroconversion post injection | 21 days after two inoculations
  * Seroconvertion is defined as: prevaccination Hemagglutination-inhibition test (HI) antibody titer ≤1:10 and postvaccination HI antibody titer ≥1:40, or prevaccination HI antibody titer ≥1:10 and a postvaccination increase by a factor of four or more.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing.
Number of participants that presented seroprotection post injection | 21 days after two inoculations
  * Seroprotection is defined as postvaccination Hemagglutination-inhibition test (HI) antibody titer ≥ 1:40.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing.
Geometric mean of Hemagglutination-inhibition titre post first study injection | 21 days after two inoculations
  * Geometric mean of Hemagglutination-inhibition test titre will be calculated for the different groups of participants post first study injection.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ze Chen, PhD, Principal Investigator — Shanghai Institute Of Biological Products
Locations (1):
- Suiping Center for Disease Control and Prevention, Zhumadian, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03369808/Prot_SAP_000.pdf